CLINICAL TRIAL: NCT02221245
Title: Interrogation of Wnt, Notch, and Hedgehog Activity in Chemonaive Tumors Collected During the Staging Ultrasound Endoscopies of Patients Diagnosed With Esophageal Cancer
Brief Title: Wnt, Notch and Hedgehog Activity in Chemo-Naive Tumors Collected During Staging of Esophageal Cancer Patients
Status: Terminated | Type: Observational
Why Stopped: Study terminated due to low accrual.
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Anthony Capobianco, Professor, University of Miami
Other Study IDs: 20120959
Record Dates: First submitted 2014-08-18; First posted 2014-08-20 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Esophageal Cancer
Keywords: Esophageal cancer; Cancer Stem Cell; CSC; Wnt; Hegdehog; Notch; Signaling; Pathway; Chemo-naive
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Esophageal cancer tumor cells
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Esophageal Cancer: Tumor Biopsy via Ultrasound Endoscopy
  Interventions: Procedure: Tumor Biopsy via Ultrasound Endoscopy

INTERVENTIONS:
Procedure: Tumor Biopsy via Ultrasound Endoscopy — The staging ultrasound endoscopy is performed on patients previously diagnosed with esophageal cancer via diagnostic biopsy. The staging ultrasound identifies affected lymph nodes and depth of tumor to the esophageal wall. The tumor sampling is via a biopsy forcep (one pass to obtain 100 cells).

SUMMARY:
Cancer results when undifferentiated cells grow in an uncontrolled manner, crowding out normal cells, causing morbidity and ultimately mortality. the cancer stem cell theory suggests that most tumors undergo a process of differentiation through which a relatively rare cancer stem or progenitor cell (CSC) gives rise to more differentiated populations of cells (including transiently amplifying cells) comprising the bulk of the tumor. As a result of this cellular diversity, one or more cells within the tumor are likely to be resistant to therapy. Among cells resistant to a given therapy, only CSCs can repopulate the tumor. A key feature of this resistant subset of CSCs is that they repopulate a tumor resistant to the original intervention. The cellular programs driving the uncontrolled proliferation of many solid tumors result from aberrant activity of Wnt, Shh, and/or Notch signaling pathways in esc. Thus, therapies that down-regulate the activity of these fundamental pathways in CSCs will be effective in the treatment of cancer. The investigator's research program focuses on the elucidation of signaling mechanisms, control of cellular processes and discovery of small molecules that selectively target Wnt, Shh, and Notch signaling pathways that are fundamental to CSCs. Our preliminary results identified a novel Notch associated protein NACK that functions as a transcriptional co-activator of Notch. Moreover, Nack is expressed in human solid tumors and is required for cell survival and tumor growth in notch -dependent tumor cells.

The investigator's aim is to further interrogate the link between Notch and Nack.

Specific Aims:

* Identify and isolate the cancer stem cell populations from primary chemo naive esophageal tumor samples.
* Interrogate the status of the Notch,( the link between Notch and Nack), Wnt and Hedghog pathways in the chemo naive esophageal tumor as well as in specific cell populations, such as the CSC.
* Determine the degree of cross-talk between these pathways and which of these pathways is essential for the self renewal properties and tumorigenic properties of the esc population.
* Identify critical targets for therapeutic intervention in CSC populations.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with an esophageal cancer and scheduled for a standard of care endoscopic ultrasound.
* Patient must sign a consent to be a participant in this protocol.

Exclusion Criteria:

* Patients not diagnosed with an esophageal cancer.
* Patients that have undergone a previous staging endoscopic ultrasound.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with esophageal cancer
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2013-04-05 (Actual); Primary Completion 2018-11-07 (Actual); Study Completion 2018-11-07 (Actual)

PRIMARY OUTCOMES:
Percentage of samples with identifiable Notch, Wnt and Hedghog pathways in the chemo naive esophageal tumor as well as in cancer stem cell populations (CSC). | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Capobianco, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States